CLINICAL TRIAL: NCT07053618
Title: Interventional Left Ventricular Assist System for PCI in CHIP Patients: a Prospective, Multicenter, Noninferiority Randomized Controlled Trial
Brief Title: Interventional Left Ventricular Assist System for PCI in CHIP Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Hengruihongyuan Medical Technology Co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVAD2.0
Record Dates: First submitted 2025-06-23; First posted 2025-07-08 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: High-Risk Percutaneous Coronary Intervention (High-risk PCI); Left Ventricular Assist Devices

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VADLINK (Experimental): The VADLINK percutaneous left ventricular assist system will offer intraoperative hemodynamic support during high-risk PCI procedures.
  Interventions: Device: Implantation of the VADLINK Percutaneous Left Ventricular Assist Device
- V-A ECMO (Active Comparator): The VA-ECMO offers intraoperative hemodynamic support during high-risk PCI procedures.
  Interventions: Device: VA-ECMO

INTERVENTIONS:
Device: Implantation of the VADLINK Percutaneous Left Ventricular Assist Device — To implant VADLINK percutaneous left ventricular assist device during percutaneous coronary intervention (PCI).
  Arms: VADLINK
Device: VA-ECMO — Received venous arterial extracorporeal membrane oxygenation (VA-ECMO) during PCI.
  Arms: V-A ECMO

SUMMARY:
Mechanical circulatory support (MCS) is a life-sustaining therapy first introduced in the 1950s. After six decades of development, it now serves as a critical bridge therapy for patients with acute cardiac events and end-stage heart failure. Percutaneous mechanical circulatory support (pMCS), a key MCS modality, has advanced rapidly in recent years.

In China, pMCS adoption has accelerated significantly, evidenced by year-over-year growth in both specialized centers and clinical cases, alongside continuous technological refinement.

Common pMCS devices include: Intra-Aortic Balloon Pump (IABP), Axial flow pump systems (e.g., Impella®), Extracorporeal Membrane Oxygenation (ECMO). However, no randomized study has compared Impella with VA-ECMO in CHIP patients.

The aim of the study is to evaluate the effectiveness and safety of interventional left ventricular assist system (VADLINK) compared to the VA-ECMO in providing circulatory support for complicated and high-risk patient with indications for PCI.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-90 2. The investigator assesses that the subject requires coronary revascularization, but CABG (Coronary Artery Bypass Grafting) is considered high-risk or the subject refuses CABG. The investigator believes the subject may benefit from PCI (Percutaneous Coronary Intervention).

3. Left ventricular ejection fraction (LVEF) ≤ 35%. 4. Coronary angiography (CAG) or coronary computed tomography angiography (CTA) shows any of the following conditions:

1. Unprotected left main (LM) coronary artery disease (coronary stenosis ≥ 50%).
2. A last remaining patent coronary artery (the anterior descending artery (LAD) and/or its branches, the circumflex artery (LCX) and/or its branches, and the right coronary artery (RCA) and/or its branches).
3. Saphenous vein graft (SVG) vascular lesions.
4. Severely calcification, tortuosity.
5. Multivessel disease (two or more) combined with chronic total occlusion (CTO).
6. Three-vessel disease. Three-vessel disease is defined as significant stenosis (≥ 70%) in at least one segment of all three major epicardial coronary artery territories: the left anterior descending artery (LAD) and/or its branches, the left circumflex artery (LCX) and/or its branches, and the right coronary artery (RCA) and/or its branches. In a left-dominant coronary system, lesions in the proximal segments of the LAD and LCX are also considered three-vessel disease.

5. Patients who are able to give informed consent and complete the follow-up.

Exclusion Criteria:

1. Cardiogenic shock (CS) within 7 days (Cardiogenic shock: Sustained SBP <90 mmHg for ≥30 min or requiring supportive measures to maintain SBP >90 mmHg and end-organ hypoperfusion (urine output <30 ml/h or cool extremities).
2. STEMI or CK-MB did not return to the normal range within 24 hours.
3. Cardiac arrest with cardiopulmonary resuscitation within 24 hours.
4. Left ventricular mural thrombus.
5. After aortic valve replacement surgery (mechanical, bioprosthetic).
6. Having used or using ECMO or pVAD (percutaneous ventricular assist device) within 7 days.
7. Moderate to severe aortic stenosis, moderate to severe aortic valve insufficiency.
8. Atrial septal or ventricular septal defects (including post-infarction VSD), or post-myocardial infarction Free-Wall Rupture, or papillary muscle rupture.
9. Severe right heart failure or severe tricuspid valve insufficiency.
10. Disease or abnormality of the aorta that interferes with the procedure, including Marfan syndrome, coarctation of aortic, aortic aneurysm, severe tortuosity or calcification of the aorta.
11. Severe peripheral arterial stenosis or occlusive lesions.
12. Uncorrectable moderate or severe anemia prior to the procedure (hemoglobin <90 g/L). Abnormal coagulation function (routine blood test indicates platelet count less than 75×109/L, INR ≥2.0, or fibrinogen ≤1.5 g/L).
13. Known contraindications to heparin, contrast agents, or study-required medications (e.g., aspirin, clopidogrel); history of Heparin-induced thrombocytopenia.
14. Active hemorrhage within 1 month.
15. History of stroke or TIA or permanent neurologic deficits within one month prior to the procedure.
16. Renal dysfunction: subject on dialysis or serum creatinine ≥4 mg/dL (353.6 µmol/L) within 7 days.
17. Liver dysfunction: liver AST, ALT and bilirubin >3 times the upper limit of normal within 7 days.
18. Presence or suspected presence of infective endocarditis or systemic infection.
19. Women who are pregnant, breastfeeding, or planning pregnancy during the trial.
20. Participation in another drug or medical device clinical trial.
21. Other conditions deemed by the investigator as unsuitable for participation in this trial.

    -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
30-day Major Adverse Events (MAE) rate | From enrollment to 30 ±7 days after PCI surgery
  Occurrence of a major adverse event (MAE) up to 30 days post-implantation. Major adverse event is a composite endpoint, defined as all-cause death, stroke, myocardial infarction, Unplanned percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG), cardiovascular hospitalization, MCS-ARC defined bleeding types 3, 4, or 5, acute kidney injury, serious device-related adverse events, cardiopulmonary resuscitation or ventricular arrhythmias after electrical cardioversion.

SECONDARY OUTCOMES:
The MACCE rate | 30, 90 days
  Incidence of Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) within 30 or 90 days after surgery.
Transfusion rate | 30 days
  Transfusion rate within 30 days after surgery.
Mean units transfused | 30 days
  Mean Number of Blood Units Transfused within 30 Days Postoperatively.
Incidence of hemodynamic instability | 30 days
  Incidence of hemodynamic instability within 30 days device implantation.
90-day Major Adverse Events (MAE) rate | 90 days
Incidence of device-related adverse events | Implant up through 90 days
Incidence of device-related serious adverse events | Implant up through 90 days
Incidence of adverse events | Implant up through 90 days
Serious adverse event incidence rate | Implant up through 90 days
Incidence of device defects | Periprocedural

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Zhongshan Hospital Affiliated to Xiamen University, Xiamen, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - People's Hospital of Hunan Province, Changsha, Hunan
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The People's Hospital of Liaoning Province, Shenyang, Liaining
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No